CLINICAL TRIAL: NCT01840098
Title: Leucine and Beta-hydroxy-beta-methylbutyrate (HMB) as Anabolic Nutrients After 36 Hours of Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Nikolaj Fibiger Rittig, MD (medical graduate) and Ph.d.-student, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-63-13
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Fasting; Metabolism; Nutrition Support
MeSH Terms: conditions — Fasting | interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (Active Comparator): Isocaloric carbohydrate drink
  Interventions: Dietary Supplement: Control/carbohydrate; Behavioral: 36 hour fasting
- low leucine content drink (Active Comparator): A soy protein drink
  Interventions: Dietary Supplement: low leucine content drink; Behavioral: 36 hour fasting
- high content of leucine drink (Active Comparator): A whey protein drink
  Interventions: Dietary Supplement: high leucine content drink; Behavioral: 36 hour fasting
- low leucine content + HMB drink (Active Comparator): Soy protein drink added HMB
  Interventions: Dietary Supplement: low leucine + HMB drink; Behavioral: 36 hour fasting

INTERVENTIONS:
Dietary Supplement: low leucine content drink
  Arms: low leucine content drink
Dietary Supplement: high leucine content drink
  Arms: high content of leucine drink
Dietary Supplement: low leucine + HMB drink
  Arms: low leucine content + HMB drink
Dietary Supplement: Control/carbohydrate
  Arms: control
Behavioral: 36 hour fasting

SUMMARY:
The purpose of this study is to investigate metabolic effects of 3 different nutritional compounds.

Fasting (36 hours) creates a catabolic state that is comparable with the catabolic state seen in acute illness.

This study is a randomized, placebo cross-over study investigating 8 healthy men on 4 separated days (at least 3 weeks between trials).

* High leucine content drink
* Low leucine content drink
* Low leucine content drink + HMB
* Carbohydrate (isocaloric)

The investigators hypothesize that these nutritional supplements may counteract catabolic processes in different ways and degrees.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* 20<BMI<30
* Age > 20 years old
* Written consent before starting the study

Exclusion Criteria:

* Allergy for soya products ore egg
* Diabetes
* Epilepsy
* Infection
* Immune defects
* Heart disease
* Dysregulated hypertension
* Participating in other trials using radioactive tracers or x-rays the last year.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Protein metabolism after 36 hours fasting receiving different nutritional supplements. | 3 control period followed by 4 hours of nutritional drink intake
  Protein metabolism is measured with amino acid tracer techniques comparing marked amino acids from blood samples. Muscle and fat biopsies are obtained for signaling analysis. Indirect calorimetry measurements are used to compare metabolism in the control period and during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine and Endocrinology, Aarhus Universitetshospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Pedersen MGB, Lauritzen ES, Svart MV, Stoy J, Sondergaard E, Thomsen HH, Kampmann U, Bjerre M, Jessen N, Moller N, Rittig N. Nutrient sensing: LEAP2 concentration in response to fasting, glucose, lactate, and beta-hydroxybutyrate in healthy young males. Am J Clin Nutr. 2023 Dec;118(6):1091-1098. doi: 10.1016/j.ajcnut.2023.10.007. Epub 2023 Oct 14. PMID 37844838
- [Derived] Rittig N, Bach E, Thomsen HH, Moller AB, Hansen J, Johannsen M, Jensen E, Serena A, Jorgensen JO, Richelsen B, Jessen N, Moller N. Anabolic effects of leucine-rich whey protein, carbohydrate, and soy protein with and without beta-hydroxy-beta-methylbutyrate (HMB) during fasting-induced catabolism: A human randomized crossover trial. Clin Nutr. 2017 Jun;36(3):697-705. doi: 10.1016/j.clnu.2016.05.004. Epub 2016 May 25. PMID 27265181